CLINICAL TRIAL: NCT02437786
Title: Molecular and Cellular Mechanism in Rhinitis Allergic Patients Treated With GRAZAX®
Acronym: GT-20
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GT-20
Record Dates: First submitted 2015-01-05; First posted 2015-05-08 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Allergic Rhinoconjunctivitis
MeSH Terms: interventions — Grazax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GRAZAX (Experimental): GRAZAX
  Interventions: Drug: GRAZAX

INTERVENTIONS:
Drug: GRAZAX — GRAZAX

SUMMARY:
The specific clinical trial is a part in which ALK- Abelló will directly work to explore human immunological mechanisms of SIT (observed after GRAZAX treatment).

DETAILED DESCRIPTION:
The main idea of the project was to address the study of some of the most important inflammatory diseases (psoriasis, rheumatoid arthritis, lupus, rhinitis/asthma… ) with the aim of identifying novel inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before entering the trial.
* Male and female 18-65 years of age.
* A clinical history of relevant rhinitis or rhinoconjunctivitis (with/without concurrent asthma) to grass pollen of at least one year prior to trial entry.
* Documented positive specific IgE against grass pollen (IgE ≥ Class 2) into the 5 previous years.
* Positive Skin Prick Test response (wheal diameter ≥ 3 mm) to Phleum pratense.
* Negative pregnancy test for childbearing potential females.
* Willing and able to comply with the trial protocol regimen.

Exclusion Criteria:

* Previous treatment by immunotherapy with grass allergen extracts.
* A clinical history of symptomatic perennial allergic rhinitis or asthma.
* Patients with contraindications for immunotherapy as established by the IT subcommittee of the EAACI or in the Summary of Products Characteristics of GRAZAX®.
* Positive pregnancy test (in fertile females).
* Being immediate family of the investigator or trial staff.
* A mental condition rendering the subject unable to understand the nature, scope and possible consequences of the trial, and/or evidence of an uncooperative attitude.
* Unlikely to be able to complete the trial, for any reason, or likely to move, or travel for extended periods of time during the trial period.
* Use of an investigational drug within 30 days or 5 half-lives, whichever is longest, prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in immunological markers (composite) measured in grass allergic subjects during treatment with Grazax® | 5 years

SECONDARY OUTCOMES:
Number of participants with IMP related adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: CARLOS BLANCO, PhD, Principal Investigator — HOSPITAL UNIVERSITARIO DE LA PRINCESA MADRID
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Suarez-Fueyo A, Ramos T, Galan A, Jimeno L, Wurtzen PA, Marin A, de Frutos C, Blanco C, Carrera AC, Barber D, Varona R. Grass tablet sublingual immunotherapy downregulates the TH2 cytokine response followed by regulatory T-cell generation. J Allergy Clin Immunol. 2014 Jan;133(1):130-8.e1-2. doi: 10.1016/j.jaci.2013.09.043. Epub 2013 Nov 28. PMID 24290282